CLINICAL TRIAL: NCT07182682
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Evaluate the Anti-Tumor Efficacy and Safety of Sunvozertinib Versus Placebo as Adjuvant Therapy in Patients With Stage IB-IIIA Non-Small Cell Lung Cancer Harboring EGFR Exon 20 Insertion Mutations or PACC Mutations After Radical Surgery (WU-KONG16)
Brief Title: A Phase 3 Study of Sunvozertinib Versus Placebo as Adjuvant Therapy in Patients With Early-Stage Non-Small Cell Lung Cancer Harboring EGFR Exon 20 Insertion Mutations or PACC Mutations After Radical Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dizal (Jiangsu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dizal Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DZ2025E0001
Record Dates: First submitted 2025-09-03; First posted 2025-09-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sunvozertinib, 200 mg orally, once daily (Experimental)
  Interventions: Drug: sunvozertinib
- Matching placebo, 200 mg orally, once daily (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: sunvozertinib — Participants will receive oral administration of sunvozertinib 200 mg QD following randomization, with each treatment cycle defined as 21 days, until meeting any treatment discontinuation criteria (i.e, objective disease recurrence, intolerable adverse event [AE], completion of 3-year [156-week] treatment period, study termination, death, treatment or study withdrawal by participants, whichever occurs first).
  Arms: Sunvozertinib, 200 mg orally, once daily
Drug: Matching Placebo — Participants will receive oral administration of placebo 200 mg QD following randomization, with each treatment cycle defined as 21 days, until meeting any treatment discontinuation criteria (i.e, objective disease recurrence, intolerable adverse event [AE], completion of 3-year [156-week] treatment period, study termination, death, treatment or study withdrawal by participants, whichever occurs first).
  Arms: Matching placebo, 200 mg orally, once daily

SUMMARY:
To assess the efficacy and safety of sunvozertinib versus placebo as adjuvant therapy in patients with stage IB-IIIA non-small cell lung cancer (NSCLC) harboring epidermal growth factor receptor (EGFR) exon 20 insertion mutations (exon20ins) or P-loop and αC-helix compression (PACC) mutations, who have had radical surgery, regardless of adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a signed and dated informed consent form (ICF) prior to any study specific procedures, sampling, and analyses.
2. Aged at least 18 years old at the time of ICF signature.
3. Complete resection (R0) of the primary tumor and histologically confirmed diagnosis of NSCLC (participants with tumor histology indicative of neuroendocrine carcinoma, sarcomatoid carcinoma, or small cell lung cancer should be excluded).

   * Complete surgical resection of the primary NSCLC is mandatory. All gross lesions must be completely resected to achieve microscopically negative margins. Hilar and mediastinal lymph node dissection should be performed per clinical guidelines.
   * Acceptable surgery type: lobectomy, sleeve lobectomy, bilobectomy, or pneumonectomy.
   * Acceptable surgery approach: thoracotomy or thoracoscopic surgery.
4. Participants must have NSCLC classified post-operatively as stage IB, II, or IIIA according to the AJCC TNM staging 9.0th edition.
5. Have documented EGFR exon20ins (Cohort 1) or EGFR PACC mutations (Cohort 2) from a local Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory (or equivalent).

   • Common EGFR PACC mutations include, but not limited to, L718Q, G719X, S768I, L747P/S, V769L, E709_T710delinsD, L792H, and T854I.
6. Participants must provide sufficient tumor tissue samples for confirmation of EGFR mutations by the sponsor designated central laboratory.
7. ECOG performance status is 0 or 1.
8. Participants must recover from prior lung surgery and systemic therapy (e.g., neoadjuvant therapy and/or adjuvant chemotherapy) without Grade 1 or higher AEs (except alopecia of any grade and ≤ Grade 2 platinum-associated neuropathy) at randomization.

   * Participants who have not previously received adjuvant chemotherapy should be randomized as early as 4 weeks and within 10 weeks after the radical surgery.
   * Participants who have previously received adjuvant chemotherapy can be randomized within 2 - 10 weeks of completion of adjuvant chemotherapy with a maximum interval of no more than 26 weeks from surgery to randomization. The adjuvant chemotherapy can start as early as 4 weeks after the radical surgery, in 21-day cycles, and up to 4 cycles.
9. Adequate bone marrow reservation or organ functions within 7 days prior to randomization.
10. Male participants with female partners of child-bearing potential should use barrier contraceptives (e.g., by use of condoms), during their participation in this study and for 6 months following the last dose of the study drug. Male participants must refrain from donating sperm during their participation in the study and for 6 months following the last dose of the study drug. If male participants wish to father children, they should be advised to arrange for freezing of sperm samples prior to the start of study drug.
11. Female participants of child-bearing potential should use reliable contraceptives from the time of screening until 2 months after discontinuation of study drug. Female participants should not be breast feeding and must have a negative pregnancy test (serum or urine β-human chorionic gonadotropin) prior to start dosing or must fulfil one of the following criteria at screening:

    * Post-menopausal defined as aged at least 50 years old and amenorrhea for at least 12 months following cessation of all exogenous hormonal treatment.
    * Women under 50 years old would be considered postmenopausal if they have been amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range.
    * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.

Exclusion Criteria:

1. Concurrent EGFR sensitizing mutations (L858R and/or exon 19 deletion) or other driver gene variations with available standard therapies (e.g., ALK positive).
2. Participants who have had only segmentectomies or wedge resections.
3. Participants who have received any preoperative or postoperative radiotherapy for NSCLC, or who plan to have radiotherapy during the study.
4. Participants who have received any EGFR TKIs as (neo)adjuvant therapy for NSCLC or have known pathological complete response from previous neoadjuvant therapy.
5. Participants who are receiving (or unable to stop) medications or herbs known to be strong CYP3A inducers within 2 weeks prior to randomization.
6. Previous history of interstitial lung disease (ILD), drug-induced ILD, or radiation pneumonitis requiring steroid therapy, any evidence of clinically active ILD, or immunotherapy induced pneumonitis.
7. Any serious or uncontrolled systemic disease requiring treatment, including uncontrolled hypertension, diabetes, chronic heart failure and active bleeding disorders (such as hemophilia, von Willebrand disease), etc., which in the opinion of the investigator is not suitable for participation in the trial or will affect compliance with the protocol; or active infection, including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
8. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) > 470 msec on 3 ECGs at screening
   * Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG, e.g., complete left bundle branch block, third degree heart block, and second-degree heart block, PR interval > 250 msec.
   * Any factors that increase the risk of QTc prolongation, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years old in first degree relatives or any concomitant medication known to prolong the QT interval.
   * Prior history of atrial fibrillation within 6 months of the first dose of study drug, except for those related to drug treatment and recovered.
9. Participants with a history of any malignancy, except for adequately treated non-melanoma skin cancer, carcinoma in situ or other solid tumors with >5 years since completion of anti-cancer therapy and no evidence of disease recurrence at randomization
10. Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous major bowel resection that may preclude adequate absorption of sunvozertinib.
11. Hypersensitivity to sunvozertinib, excipients of sunvozertinib, or drugs of similar chemical structure or same class.
12. Involvement in the design, planning or conduct of this study (applicable to Dizal staff or study site staff).
13. Judgment by the investigator that the participant is unlikely to comply with study procedures, restrictions or requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) by investigator assessment | Up to approximately 5 years after the first participant is randomized

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 5 years after the first participant is randomized.
DFS rate at 2, 3, and 5 years by investigator assessment | Up to approximately 5 years after the first participant is randomized.
OS rate at 2, 3 and 5 years | Up to approximately 5 years after the first participant is randomized.
Incidence of adverse event (AE) and serious adverse event (SAE) | Up to approximately 3 years after the first dose
The plasma concentration of sunvozertinib and its metabolite (DZ0753) | Up to approximately 3 years after the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Zhou, Principal Investigator — Shanghai East Hospital; Wang, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (49):
- China (49):
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital, Capital medical university, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - China-Japan Friendship hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - The Third Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital of Central South University, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Fujian Medical University Union Hospital, Fuzhou
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Cancer Hospital, Hefei
  - Jinan Central Hospital, Jinan
  - Shandong Cancer Hospital, Jinan
  - Yunnan Cancer Hospital, Kunming
  - Jiangxi Provincial People 's Hospital, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Nanjing Chest Hospital, Nanjing
  - Guangxi Medical University Cancer Hospital, Nanning
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Shanghai East Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The First Hospital of China Medical University, Shenyang
  - Shanxi Cancer hospital (Shanxi Cancer institute), Taiyuan
  - Shanxi Provincial people's hospital, Taiyuan
  - Taizhou Hospital, Zhejiang Province, Taizhou
  - Tianjin Chest Hospital, Tianjin
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Henan Cancer Hospital, Zhengzhou
  - The first affiliated hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No